CLINICAL TRIAL: NCT02862210
Title: Low-Dose Lithium for the Treatment of Behavioral Symptoms in Frontotemporal Dementia
Acronym: Lithium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Principal Investigator, Edward D Huey, MD, Assistant Professor of Psychiatry, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NYSPI 7310
Record Dates: First submitted 2016-08-07; First posted 2016-08-10 (Estimated); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Frontotemporal Dementia (FTD)
Keywords: Lithium; Lithium Carbonate
MeSH Terms: conditions — Frontotemporal Dementia | interventions — Lithium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lithium carbonate (Experimental): Lithium will be prescribed starting at 150 mg/day, with subsequent dose titration to 300, 450, and 600 mg/day as tolerated according to side effects and blood lithium level.
  Interventions: Drug: Lithium Carbonate
- Placebo (Placebo Comparator): Placebo will be prescribed starting at 1 pill per day, with subsequent dose titration to 2,3, and 4 pills per day as tolerated by sham blood lithium levels provided by an unblinded study team member.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium Carbonate — Lithium will be prescribed starting at 150 mg/day, with subsequent dose titration to 300, 450, and 600 mg/day as tolerated according to side effects and blood lithium level.
  Other Names: Lithobid
  Arms: Lithium carbonate
Drug: Placebo — Placebo will be prescribed starting at 1 pill per day, with subsequent dose titration to 2,3, and 4 pills per day as tolerated by sham blood lithium levels.
  Arms: Placebo

SUMMARY:
Frontotemporal dementia (FTD) is a progressive neurodegenerative illness that affects the frontal and anterior temporal lobes of the brain. Changes in behavior, including agitation, aggression, and repetitive behaviors, are common symptoms in FTD. The investigators currently do not have good medications to treat these symptoms in FTD, and the medications the investigators use often have side effects. In this project, the investigators will test the use of low-dose lithium, compared to a placebo pill, for the treatment of behavioral symptoms in FTD. Lithium greatly reduces the behavioral symptoms of bipolar disorder, and many have found low-dose lithium to be well-tolerated in patients with dementia. Lithium appears to inhibit the creation of a protein involved in many cases of FTD called tau.

DETAILED DESCRIPTION:
Behavioral symptoms of Frontotemporal dementia (FTD), including agitation, aggression, and inappropriate repetitive behaviors are common, distressing to patients and caregivers, often lead to institutionalization, and can be very difficult and expensive to treat. There is a dearth of medication for treating these symptoms in FTD. Typically, antidepressants and antipsychotic medications are prescribed - which low efficacy and, with the latter class, carry serious adverse effects such as parkinsonism and increased cardiovascular-related mortality. The investigators propose a study of the efficacy of lithium carbonate compared to placebo in the treatment of agitation, aggression, and inappropriate repetitive behaviors in 60 patients with FTD in a randomized, double-blind, two-arm parallel 12-week trial. Lithium is a highly effective treatment for mania and symptoms of agitation or aggression in bipolar disorder. It also inhibits tau aggregation and phosphorylation, leading to considerable interest in its use as a disease-modifying treatment for tauopathies such as FTD and Alzheimer's disease. Unfortunately, earlier trials using typical doses (i.e., doses prescribed for treatment of bipolar disorder) showed high incidence of serious adverse effects (including confusion and delirium). For this proposed study the investigators will: 1) use lower doses and lower target serum concentrations than have preceding trials (shown in preliminary data from a Columbia study and data from other labs to be well-tolerated) and 2) target behavioral symptoms rather than cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-85
* A diagnosis of behavioral variant FTD (bv-FTD) or semantic variant Primary Progressive Aphasia (sv-PPA, which is generally accompanied by a behavioral syndrome), or agrammatic/non-fluent Primary Progressive Aphasia (nfv-PPA) with behavioral symptoms
* Neuropsychiatric Inventory (NPI) agitation/aggression subscale score ≥4 or disinhibition subscale score ≥ 4 or repetitive behavior subscale ≥ 4 or total score ≥ 6. On each subscale, a score higher than 4 represents moderate to severe symptoms
* Folstein Mini-Mental State Examination (MMSE) score 5-26/30
* An study partner (usually a family member) is required to provide information during interviews about the patient
* Capacity to consent. Subjects without capacity to consent must have capacity to appoint a surrogate
* Structural MRI or CT scan after symptom onset

Exclusion Criteria:

* Medical contraindication or history of intolerability to lithium, falls in the last month, current abnormal thyroid functions (T3, T4 or thyroid stimulating hormone (TSH); treated hypothyroidism with normal thyroid function tests will not lead to exclusion), creatinine level > 1.5 mg/100 ml or glomerular filtration rate < 44 ml/min/1.73m2 will also lead to exclusion
* The diagnosis of bipolar disorder or schizophrenia or schizoaffective disorder
* Alcohol or substance use disorder in the prior 6 months
* Current diagnosis of other major neurological disorder, e.g., Alzheimer's Disease (AD), stroke with residual clinical deficits, multiple sclerosis, Parkinson's disease. Subjects with MRI or CT evidence of cerebrovascular disease but without clinical signs of stroke will be included
* Sitting blood pressure > 150/90 mm Hg, unstable cardiac disease, severe or unstable medical illness
* Use of medications, including diuretics, known to have adverse effects when combined with lithium. Use of antipsychotic medications will be permitted
* Current major depression or suicidality or dangerous behavior with risk of harm to self and others
* Corrected QT interval (QTc) interval > 460 ms at the time of baseline electrocardiogram (EKG)
* Woman of child-bearing potential

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2022-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Huey, MD, Principal Investigator — Brown University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 17 participants signed a consent form. One participant was a screen failure, resulting in randomization of 16 participants.
Period: Overall Study
Arm/Group | Lithium Carbonate | Placebo
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lithium Carbonate | Placebo | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Customized [Count of Participants; unit: Participants]
  40-55 years | 2 | 3 | 5
  56-65 years | 5 | 2 | 7
  66-75 years | 2 | 2 | 4
  76-85 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Agitation and Aggression as Measured by the Neuropsychiatric Inventory Scale (NPI)
Description: The NPI is a scale designed to assess behavioral changes due to neurological illness. It uses a standardized caregiver interview to rate patient symptoms in a variety of domains, including "Agitation/Aggression." Each domain includes a number of questions about potential specific symptoms, and then asks the caregiver to rate symptom frequency (1, occasionally, to 4, very frequently) as well as symptom severity (1, mild, to 3, severe). Scores range from from 0-12, with 0 being no symptoms and 12 being very frequent and severe symptoms. The study aims to test the effect of lithium on agitation/aggression as compared to placebo by testing whether participants taking lithium show a greater reduction in their NPI "Agitation/Aggression" domain score over the course of the trial.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
score on a scale | 7.14 (1.1) | 5.75 (1.28)

2. Secondary Outcome: Number of Responders in the Lithium and Placebo Groups
Description: Responder defined as a 30% decrease in NPI core score (sum of domain scores for "Agitation/Aggression" and "Aberrant Motor Behavior") plus a Clinical Global Impression (CGI) Change score of much improved or very much improved (CGI based on these behavioral symptoms only).
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
participants | 0 | 0

3. Other Pre Specified Outcome: Change in Motor Symptoms as Measured by the NPI
Description: NPI domain "Aberrant Motor Behaviors" will be observed to test the effect of lithium on repetitive behaviors as compared to placebo, by examining whether participants taking lithium show a greater reduction in their "Aberrant Motor Behaviors" NPI domain score. Scores range from from 0-12, with 0 being no symptoms and 12 being very frequent and severe symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
score on a scale | 6.83 (0.95) | 8.8 (1.23)

4. Other Pre Specified Outcome: Presence of Adverse Events as Measured by the Treatment Emergent Symptoms Scale (TESS)
Description: The tolerability of low-dose lithium by assessing emergent side effects over the course of the 12-week trial will be assessed. The side effects will be captured with TESS in which 30 symptoms are rated either "Absent," "Mild," "Moderate," or "Severe." The change in TESS score from baseline to week 12 will be observed. Total scores range from 0 to 96 with a higher score indicating a worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
score on a scale | 31.1 (0.55) | 31 (0.66)

5. Other Pre Specified Outcome: The Relationship Between Changes in Brain-derived Neurotropic Factor (BDNF) Serum Levels and Changes in NPI "Agitation/Aggression" Score
Description: The baseline serum BDNF levels as a potential baseline predictor of lithium treatment response and an increase from pre to post-treatment BDNF levels as a potential biomarker correlate of improvement in symptoms (as measured by the NPI) will be explored. The mean change of NPI "Agitation/Aggression" score as a function of BDNF level change from baseline to 12 weeks will be reported. Scores range from from 0-12, with 0 being no symptoms and 12 being very frequent and severe symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
score on a scale | 0.71 (1.91) | -1.6 (2.11)

6. Other Pre Specified Outcome: The Relationship Between Changes in Brain-derived Neurotropic Factor (BDNF) Serum Levels and Changes in NPI "Aberrant Motor Behavior" Score
Description: The baseline serum BDNF levels as a potential baseline predictor of lithium treatment response and an increase from pre to post-treatment BDNF levels as a potential biomarker correlate of improvement in symptoms (as measured by the NPI) will be explored. Aberrant motor behavior is characterized by repetitive movements and inability to sit still. The mean change of NPI Aberrant Motor Behavior score as a function of BDNF level change from baseline to 12 weeks will be reported. Scores range from from 0-12, with 0 being no symptoms and 12 being very frequent and severe symptoms.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lithium Carbonate | Placebo
Number analyzed (Participants) | 9 | 7
score on a scale | 0.4 (11.33) | 0.4 (1.83)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Lithium Carbonate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lithium Carbonate (N=9) | Placebo (N=7)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/10/NCT02862210/Prot_SAP_000.pdf